CLINICAL TRIAL: NCT00518596
Title: Prevention of Infection in Indian Neonates - Phase II Probiotics Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); All India Institute of Medical Sciences (Other); TN Medical College, Mumbai (Other); Department of Health and Family Welfare, Orissa (Other); SCB Medical College, Cuttack (Other); Capital Hospital, Bhubaneswar (Other); Ispat General Hospital, Rourkela (Other); Kalinga Hospital, Bhubaneswar (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GN 07 Phase II; U01HD040574 (NIH); R01HD053719 (NIH)
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Sepsis
Keywords: Neonatal; Sepsis; Global Network; Probiotics; India; International; Maternal and child health
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Probiotic Arm (Experimental): Newborn infants' ≥ 35 weeks of gestation and ≥1800g, given L. plantarum preparations orally once a day starting on day 1, 2, or 3 of life and continuing for seven days thereafter.
  Interventions: Dietary Supplement: Probiotic supplementation (Lactobacillus plantarum)
- Control Arm (Placebo Comparator): Newborn infants' ≥ 35 weeks of gestation and ≥1800g, receiving placebo preparations (a control solution of sterile 2.0 cc 5% dextrose-saline)orally once a day starting on day 1, 2, or 3 of life and continuing for seven days thereafter.
  Interventions: Dietary Supplement: Probiotic supplementation (Lactobacillus plantarum)

INTERVENTIONS:
Dietary Supplement: Probiotic supplementation (Lactobacillus plantarum) — GastroPlan capsules from a single lot will be used. The intervention consists of L. plantarum reconstituted in sterile 2.0 cc of 5% dextrose-saline, administered orally using an opaque-amber syringe.
  Other Names: Gastroplan

SUMMARY:
India, with one of the world's largest populations, continues to struggle with extremely high infant and neonatal mortality rates. Neonatal infection (sepsis) now accounts for 50 percent of deaths among community-born (and 20 percent of mortality among hospital-born) infants. This study is the first phase of a multi-phase project investigating interventions to prevent neonatal infection in India.

DETAILED DESCRIPTION:
Phase II is a hospital based intervention (n = 297 infants) measuring the colonizing ability, safety, and tolerance of a probiotic supplement, Lactobacillus plantarum in the neonatal gut. Newborn infants ≥ 35 weeks of gestation will be randomized to receive either L. plantarum preparations (containing 109 organisms) or placebo preparations orally once a day for the first 7 days of life. The final stage of the project will be a community-based randomized double-blind placebo-controlled trial of L. plantarum enrolling over 8,000 newborns to examine the efficacy of probiotic supplementation in reducing neonatal infection in Indian neonates.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥ 35 weeks and ≥1800g born in the hospital
* Infants > 12 hours and < 72 hours of age at enrollment
* Infants likely to be hospitalized for 5-7 days without antibiotic treatment
* Informed consent by one parent or guardian
* Infants begun breastfeeding

Exclusion Criteria:

* Antibiotic therapy prior to enrollment
* Evidence or suspicion of clinical sepsis before randomization
* Inability (as determined by the physician) to tolerate oral feeding of study supplement
* Presence of major congenital anomalies
* Infant's home is >30km away from hospital A major congenital anomaly is defined as any malformation that is felt to be life-threatening or that requires surgical intervention. If the medical officer is uncertain whether an anomaly is life-threatening, he/she should not enroll the infant.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2005-07; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Colonizing ability of L. plantarum in Indian neonates after 5-7 days of administration. | 28 days
Clinical safety (including sepsis and death) and tolerance of a daily administration of oral L. plantarum probiotic supplement when used in healthy full-term neonates. | 28 days
Changes in stool microfloral patterns with 5-7 day administration of L. plantarum supplement.

SECONDARY OUTCOMES:
Feasibility of the future community study (consent and retention rates, completeness of stool sampling, ability to complete the study in the home for infants discharged early).

CONTACTS AND LOCATIONS:
Overall Officials: Pinaki Panigrahi, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (3):
- India (3):
  - Capital Hospital, Bhubaneswar, Odisha
  - Kalinga Hospital, Bhubaneswar, Odisha
  - Ispat General Hospital, Rourkela, Odisha

REFERENCES:
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org
- See also: RTI International — http://www.rti.org